CLINICAL TRIAL: NCT05386082
Title: Development of a Standardized Set of Core Metrics to Assess the Quality of Anesthesia, Perioperative Care, and Acute Pain Management in Canada: Scoping Review and Multidisciplinary Consensus Delphi Study
Brief Title: Anesthesia Core Quality Metrics Consensus Delphi Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Matthias Görges, PhD, Associate Professor, University of British Columbia
Other Study IDs: H22-00519
Record Dates: First submitted 2022-05-05; First posted 2022-05-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; Consensus Development
Keywords: Metrics; Perioperative care; Quality of anesthesia; Outcomes; Delphi

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: Study participants
  Interventions: Other: Modified Delphi process

INTERVENTIONS:
Other: Modified Delphi process — The study involves a brief demographics survey and Delphi process, i.e. three rounds of information and surveys, in which participants will be asked to score/rank potential metrics.

SUMMARY:
To develop a ranked list of up to 20 metrics, which can be used to evaluate the quality of anesthesia, perioperative care, and acute pain management for adult inpatient non-cardiac surgical patients for use in quality improvement and quality assurance, research, and continuing medical education in the Canadian care context.

DETAILED DESCRIPTION:
Background: Improving anesthesiology care and perioperative outcomes is a growing field encompassing quality improvement and quality assurance, research, and continuing medical education. Multiple consensus initiatives have standardized perioperative endpoints. However, no standard set of metrics exist to evaluate the quality of Canadian anesthesiology care delivery.

Objective: Develop a ranked list of up to 20 metrics, which can be used to evaluate the quality of anesthesia, perioperative care, and acute pain management for adult inpatient non-cardiac surgical patients for use in quality improvement and quality assurance, research, and continuing medical education in the Canadian care context.

Methods: First, the steering committee will conduct a scoping review of the literature to identify candidate metrics, according to Preferred Reporting Items for Systematic Reviews and Meta-Analyses extension for scoping reviews (PRISMA-ScR) and Joanna Briggs Institute methodology for scoping reviews. Metrics will include patient-reported outcome and patient-reported experience measures, quality and safety indicators, process metrics, and Canadian Anesthesiologists' Society recommended practice standards. The search strategy will include English-language articles published or in use within the past seven years (2015/Jan-2022/March) in 1) MEDLINE, Embase, CINAHL, Web of Science, and Cochrane Database of Systematic Reviews, 2) grey literature, including guidelines, and 3) existing evaluation metrics used by Canadian departments for quality assurance and improvement. Screening and data extraction will be performed by two independent reviewers using Covidence.

Next, following approval from the Research Ethics Board and with written informed consent from participants, a multidisciplinary panel of anesthesiologists, people with lived surgical experience (patients, caregivers), surgeons, nurses, internal medicine and family physicians, hospital administrators, and researchers will iteratively review the list of candidate metrics using a modified Delphi process. Independent voting, using surveys over three rounds, will be used to identify the most important metrics to define the quality of anesthesia, perioperative care, and acute pain management. Additional cycles may be performed if required.

ELIGIBILITY:
Inclusion Criteria:

* Patient/family participants must have undergone a surgical experience within the past three years, and have the capacity to provide informed consent.
* All other participants must be actively practising in Canada in the disciplines they represent.

Exclusion Criteria:

- Participants with self-declared conflicts of interest with this project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators aim to recruit 77 participants with the following characteristics: a) 26 anesthesiologists, b) 26 patients and/or their family members/caregivers, c) 9 surgeons, d) 4 nurses, e) 2 physicians each from internal medicine, emergency department, family practice, family practice anesthetists, and 4 health administrators or quality improvement leads
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Ranked list of anesthesia, perioperative care, and acute pain management quality metrics | late 2022
  A ranked set of national consensus metrics for evaluating the quality of anesthesia, perioperative care, and acute pain management for adult noncardiac surgical patients that can be used for quality improvement and quality assurance, research, and continuing medical education in the Canadian care context. Metrics where >70% participants voted "definitely priority" will be marked in the publication as the core metric set.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Görges, PhD, Principal Investigator — The University of British Columbia
Locations (3):
- Canada (3):
  - BC Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- See also: Scoping review registration — https://doi.org/10.17605/OSF.IO/8BNVW

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT05386082/Prot_SAP_000.pdf